CLINICAL TRIAL: NCT02610452
Title: Assessing the Impact of Clown Therapy in a Palliative Care Unit: A Prospective, Descriptive Study
Acronym: OUPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LOCAL/2015/SB-01; 2015-A00719-40 (Other: RCB number)
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Palliative Care
Keywords: clown therapy
MeSH Terms: interventions — Laughter Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The study population (Experimental): The study population consists of adult patients treated in the Palliative Care Unit of the University Hospital of Nimes, regardless of their original condition. In 2013 the proportion of stays connected with diagnostics for cancer was 70.16%.
  Intervention: Clown therapy
  Interventions: Other: Clown therapy

INTERVENTIONS:
Other: Clown therapy — The clowns intervene by twos: a game takes place.
  1. The game requires the active presence of a number of potential players in the room (patient, family, caregivers) and takes into account body position, emotional state, the general atmosphere.
  2. The clowns initiate a game proposal: provisional staging of clown characters based on imagination/improvisation which engages a physicality and a basic emotional state.
  3. The original game proposal is adjusted according to mutual empathy with those present.
  4. The game is developed on the model of theatrical improvisation: an original creation that has "scenic" quality comparable to that of a complete representation. Improvisation time varies depending on the condition of the person, his/her desire to participate, choosing the main theme.
  5. The final stage of the game is preparing all actors for separation: restitution of roles, revisiting the paths traveled.

SUMMARY:
The main objective of this study was to assess changes in the quality of life of patients in a Palliative Care Unit via the symptoms by the Edmonton Symptom Assessment System (ESAS) before and one hour after the passage of a clown therapist .

DETAILED DESCRIPTION:
The secondary objectives of this study are to evaluate before versus after the intervention of clowns therapists:

A. Changes in the quality of life at two days after the intervention (using the ESAS).

B. The quality of life two days after the intervention via the McGill Quality of Life Questionnaire.

C. The quality of life of patients after the intervention as assessed by semi-structured interviews conducted by the department psychologist.

D. The quality of life of caregivers after the intervention as assessed by semi-structured interviews conducted by the department psychologist.

E. Employee satisfaction at the end of the intervention period in the department and after debriefing as assessed by semi-structured interviews conducted by the department psychologist.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* Patient receiving palliative care, ie with a severe and progressive disease bringing into play vital prognosis, in advanced or terminal phase
* Clinically stable patients, regardless of disease type. The existence of clinical symptoms (pain, discomfort, etc.) found at recruitment by the investigator and not affecting the mental clarity of the subject, does not justify the exclusion of the patient
* Absence of cognitive disorders; since the protocol provides a clinical interview covering in particular his/her quality of life, included patients will be able to express their feelings
* In addition, patients who have undergone this type of intervention (clown therapist) will not be excluded from this study.

Exclusion Criteria:

* The patient is participating in another study
* The patient is an adult under judicial protection
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* Patient with an inability to fill our protocol assessment scales
* Patients under treatment known to reduce the level of awareness
* Patients with major cognitive impairment
* Patients with symptoms that bring into question their level of awareness
* Patients with significant risk factors and who should benefit from personalized monitoring from the team (clinically unstable patients, emergency situations, agitated patients, dementia, etc ...).
* Patient is unable to submit to the continuity of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2016-11-12 (Actual); Study Completion 2016-11-12 (Actual)

PRIMARY OUTCOMES:
ESAS questionnaire | 1 hour before clown therapy session
  The ESAS (Edmonton Symptom Assessment System) self-administered questionnaire
ESAS questionnaire | 1 hour after clown therapy session
  The ESAS (Edmonton Symptom Assessment System) self-administered questionnaire
ESAS questionnaire | Day 2
  The ESAS (Edmonton Symptom Assessment System) self-administered questionnaire

SECONDARY OUTCOMES:
McGill Quality of Life Questionnaire | 1 hour before clown therapy session
McGill Quality of Life Questionnaire | Day 2
Semi-directed patient interview | Day 2
Semi-directed caregiver interview | Day 0
Semi-directed staff interview | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Blanchard, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France